CLINICAL TRIAL: NCT02353182
Title: An Open Label Pilot Study of Feasibility of a Dexmedetomidine-Remifentanil-Caudal Anaesthetic for Infant Lower Abdominal/Lower Extremity Surgery: The TREX Pilot Study
Brief Title: The T REX Pilot Study: a Study to Investigate the Use of an Alternative Anaesthetic in Infants.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Murdoch Childrens Research Institute (Other)
Collaborators: Baylor College of Medicine (Other); Boston Children's Hospital (Other); Oregon Health and Science University (Other); Royal Children's Hospital (Other); UMC Utrecht (Other); Children's Hospital Medical Center, Cincinnati (Other); Children's Hospital of Philadelphia (Other); Sydney Children's Hospitals Network (Other); The Cleveland Clinic (Other); Princess Margaret Hospital for Children (Other); University Hospital, Geneva (Other); Starship Children's Health (Unknown); University of Texas Southwestern Medical Center (Other); Gaslini Children's Hospital (Other); KK Women's and Children's Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 35014
Record Dates: First submitted 2015-01-26; First posted 2015-02-02 (Estimated); Last update posted 2016-10-26 (Estimated); Status verified 2016-10

CONDITIONS: Surgical Procedures, Operative
Keywords: abdominal; lower extremity
MeSH Terms: interventions — Dexmedetomidine; Remifentanil; Bupivacaine; Ropivacaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Active open label single arm (Experimental): Dexmedetomidine- remifentanil- caudal based anaesthetic for lower abdominal/lower extremity surgery.
  Dexmedetomidine (Precedex): loading dose: 1 mcg/kg over 10 minutes. Infusion: Start 1 mcg/kg/hr; titrate up or down within 50% of starting doses as needed
  Remifentanil (Ultiva): loading dose: 1 mcg/kg over 1-2 minutes. Infusion: Start at 0.2 mcg/kg/min. Titrate up or down (max 0.5 mcg/kg/min) as needed
  Caudal- Bupivacaine (Marcaine) 0.175%-0.25% or Ropivacaine (Naropin) 0.2% with dose at discretion of anaesthetist
  Interventions: Drug: Dexmedetomidine; Drug: Remifentanil; Drug: Bupivacaine; Drug: Ropivacaine

INTERVENTIONS:
Drug: Dexmedetomidine — Loading dose:1 mcg/kg over 10 minutes. Infusion: Start 1-1.5 mcg/kg/hr. Titrate up or down within 50% of starting doses as needed.
  Other Names: Precedex
Drug: Remifentanil — Loading dose: 1 mcg/kg over 1-2 minutes. Infusion: Start at 0.2-0.5 mcg/kg/min. Titrate up or down (max 0.5 mcg/kg/min) as needed.
  Other Names: Ultiva
Drug: Bupivacaine — Administered in caudal/epidural/field block: 0.175%-0.25% (dose at discretion of anaesthetist)
  Other Names: Marcaine
Drug: Ropivacaine — Administered in caudal/epidural/field block: 0.2% (dose at discretion of anaesthetist)
  Other Names: Naropin

SUMMARY:
Animal studies suggest general anaesthetics harm the developing brain. It is unclear if these findings are relevant to humans but the issue has become a major concern. Recent data have found that monkeys exposed to anaesthesia as infants grow up to have slower learning than those not exposed.

The aim of the TREX pilot study is to determine the feasibility of an alternative anaesthetic regimen for lower abdominal/lower extremity surgery in infants 1-12 months of age.

DETAILED DESCRIPTION:
Animal studies suggest general anaesthetics harm the developing brain. It is unclear if these findings are relevant to humans but the issue has become a major concern. Recent data have found that monkeys exposed to anaesthesia as infants grow up to have slower learning than those not exposed.

The aim of the TREX pilot study is to determine the feasibility of an alternative anaesthetic regimen for lower abdominal/lower extremity surgery in infants 1-12 months of age.

An alternative anaesthetic regimen comprises a dexmedetomidine-based anaesthetic, augmented with an opioid (remifentanil) and a regional nerve block (such as a caudal).

This open label prospective single arm pilot study will enrol 60 infants aged 1-12 months scheduled for lower limb, urologic, or lower abdominal surgery. After sevoflurane induction, the infants will have a caudal anaesthetic and intravenous dexmedetomidine and remifentanil.

The outcome will be need for intervention for light anaesthesia, intervention for haemodynamic changes and rate of abandoning the protocol. Recovery times will also be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Infants aged 1 to 12 months (corrected age)
* ASA I or II
* Infants undergoing lower abdominal/lower extremity surgery anticipated to be > 120 minutes in duration
* Surgery requires caudal regional nerve block

Exclusion Criteria:

* ASA III or higher
* Any contraindication to caudal analgesia
* Any contraindication to an inhalational induction with sevoflurane
* Allergies to any medication in study protocol
* Planned admission to an ICU postoperatively (except level II or III neonatal ICU)
* Planned tracheal intubation postoperatively
* Mechanical ventilation postoperatively

Ages: 1 Month to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2015-05; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Number of participants who need for intervention for light anaesthesia | 120 minutes (duration of surgery)
  Rescue treatment for light anaesthesia will be given if hypertension MAP > 80 mmHg (confirmed with repeated measure) and/or patient movement.

SECONDARY OUTCOMES:
Number of participants who need for intervention for haemodynamic changes | 120 minutes (duration of surgery)
  1. Rescue treatment for mild Hypotension will be given if MAP is between 40 mmHg and <50 mmHg (confirmed with repeated measure)
  2. Moderate Hypotension will be defined as MAP <40 mmHg
  3. Mild bradycardia will be defined as HR <100 bpm for over one minute
  4. Significant bradycardia will be defined as <70 bpm over one minute
Time to recovery after anaesthesia | Time from last dressing to: eye opening, removal of airway device, first feed, and a modified Aldrete Score of 9-10 (average 30 minutes-4 hours)
Number of participants who have respiratory complications | Start of anaesthesia until discharge from PACU (average 1-4 hours)
  Any episode of coughing, oxygen desaturation <90%, breath holding > 15 seconds
Number of participants who have pain after anaesthesia | End of surgery until discharge from PACU ( average 1-4 hours)
  FLACC (Face, Legs, Activity, Cry, Consolability) scale. The scale is scored in a range of 0-10 with 0 representing no pain.
Number of participants who require rescue analgesia in PACU | End of surgery until discharge from PACU (average 1-4 hours)
  Analgesia: morphine 0.025-0.05 mg/kg IV for analgesia; repeat 20 minutes. Analgesia thereafter as per local protocol

CONTACTS AND LOCATIONS:
Overall Officials: Andrew J Davidson, MD, Principal Investigator — Murdoch Childrens Research Institute
Locations (6):
- United States (4):
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - The University of Texas Southwestern Medical Center, Dallas, Texas
  - Texas Children's Hospital, Houston, Texas
- Royal Children's Hospital, Parkville, Victoria, Australia
- KK Women's and Children's Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No
Data will be presented as group data and no individual will be identified.